CLINICAL TRIAL: NCT02942381
Title: A Study of Hydroxychloroquine Sulfate for Reduction of Proteinuria in Patients With IgA Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Lijun Liu, Clinical Professor, Peking University First Hospital Research department, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016(1057)
Record Dates: First submitted 2016-10-14; First posted 2016-10-24 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: IgA Patients; Hydroxychloroquine
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydroxychloroquine Sulfate (Active Comparator): 200mg Bid (eGFR>60 ml/min/1.73m2), 100mg Tid (eGFR45-59 ml/min/1.73m2), 100mg Bid (eGFR 30-44 ml/min/1.73m2) and supportive treatment
  Interventions: Drug: Hydroxychloroquine Sulfate
- Placebo (Placebo Comparator): Placebo and supportive treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — 200mg Bid (eGFR>60 ml/min/1.73m2 ), 100mg Tid(eGFR45-59 ml/min/1.73m2 ), 100mg Bid(eGFR 30-44 ml/min/1.73m2 )
  Arms: Hydroxychloroquine Sulfate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators study will recruit IgA nephropathy patients with proteinuria range from 0.75 to 3.5g/d even after three-month treatment by sufficient ACEi/ARB. The patients were treated with Hydroxychloroquine 200-400mg/d according to eGFR. The proteinuria will recorded every two months and total four months. Then, the drug will be stopped for two months for observation of change of proteinuria.

DETAILED DESCRIPTION:
Immunoglobulin A (IgA) nephropathy is the most common type of primary glomerulonephritis worldwide. Several studies indicated that 6-43% of IgA nephropathy patients would develop end-stage kidney disease (ESKD) over a period of 10 years. The clinical risk factors for progression are hypertension, proteinuria, impaired renal function and histologic lesions at presentation. There is no well accepted optimal therapy for patients with IgA. Current established therapies include full RAS inhibition and optimal blood pressure control for patients with proteinuria and/or hypertension.

Hydroxychloroquine has been used for many years to treat malaria. It is also used to treat systemic lupus erythematosus, rheumatic disorders like rheumatoid arthritis and Sjögren's Syndrome. Recently, several studies found that Hydroxychloroquine could reduce the risk of ESRD in patients with lupus nephritis. The mechanism of the treatment wasn't well known so far. Some investigators found that Hydroxychloroquine increases lysosomal pH in antigen presenting cells. In inflammatory conditions, it blocks toll-like receptors on plasmacytoid dendritic cells (PDCs). Toll-like receptor 9 (TLR 9), which recognizes DNA-containing immune complexes, leads to the production of interferon and causes the dendritic cells to mature and present antigen to T cells. Hydroxychloroquine, by decreasing TLR signaling, reduces the activation of dendritic cells and the inflammatory process.

The pathogenesis of IgA nephropathy included the deposition of immune complex containing IgA in mesangium and causing local immune activation and injury to kidney. Therefore, Hydroxychloroquine might have the potential effect of anti-inflammation in patients with IgA nephropathy, reduced the proteinuria and had the renal protect effect.

The investigators study will recruit IgA nephropathy patients with proteinuria range from 0.75 to 3.5g/d even after three-month treatment by sufficient ACEi/ARB. The patients were treated with Hydroxychloroquine 200-400mg/d according to eGFR. The proteinuria will recorded every two months and total four months. Then, the drug will be stopped for two months for observation of change of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* primary IgA nephropathy
* age 18-75 years
* proteinuria range from 0.75 to 3.5g/d even after three-month treatment by sufficient ACEi/ARB
* eGFR>30ml/min/1.73m2

Exclusion Criteria:

* immune suppressive agent in recent one years
* crescent glomerulonephritis, might use immune suppressive agent
* chronic hepatic disease
* myocardial infarction
* malignant hypertension
* stroke
* malignant tumor
* retinopathy
* other contraindication of Hydroxychloroquine
* pregnancy and breastfeeding women
* life expectancy for less than 6 months
* in other clinical trials
* not suitable for the study judged by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Proteinuria （g/d） | every two months(total six months)

SECONDARY OUTCOMES:
Albuminuria and creatinine ratio(mg/g) | every two months(total six months)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Liu LJ, Yang YZ, Shi SF, Bao YF, Yang C, Zhu SN, Sui GL, Chen YQ, Lv JC, Zhang H. Effects of Hydroxychloroquine on Proteinuria in IgA Nephropathy: A Randomized Controlled Trial. Am J Kidney Dis. 2019 Jul;74(1):15-22. doi: 10.1053/j.ajkd.2019.01.026. Epub 2019 Mar 25. PMID 30922594